CLINICAL TRIAL: NCT04447768
Title: A Phase II: Venetoclax-Based Therapy for the Treatment of Fit Patients With Chronic Lymphocytic Leukemia (CLL) in the Front-Line Setting
Brief Title: The Combination of Venetoclax and Obinutuzumab in People With Chronic Lymphocytic Leukemia (CLL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-044
Record Dates: First submitted 2020-06-24; First posted 2020-06-25 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: Venetoclax; Obinutuzumab; 20-044
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — obinutuzumab; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Venetoclax and Obinutuzumab (Experimental): All patients will receive a minimum of 9 cycles (cycle = 28 days) of therapy with venetoclax and obinutuzumab during the treatment period. For patients who remain MRD positive at Cycle 9 of therapy, an additional 12 cycles of venetoclax monotherapy will be given.
  Interventions: Drug: Obinutuzumab; Drug: Venetoclax

INTERVENTIONS:
Drug: Obinutuzumab — Cycle 1, Day 1- 100 mg
  Cycle 1, Day 2 - 900 mg
  Cycle 1, Day 8 - 1000 mg
  Cycle 1, Day 15 -1000 mg
  Cycle 2, Day 1 to Cycle 6, Day 1- 1000 mg
Drug: Venetoclax — Cycle 1, Day 22 to 28 -20 mg daily
  Cycle 2, Day 1 to Day 7 -50 mg daily
  Cycle 2, Day 8 to Day 14- 100 mg daily
  Cycle 2, Day 15 to Day 21- 200 mg daily
  Cycle 2, Day 22 to Day 28 - 400 mg daily
  Cycle 3, Day 1 to end of Cycle 12-24 - 400 mg daily

SUMMARY:
This study will help researchers collect more information about how effective the combination of venetoclax and obinutuzumab is in treating CLL in people who have not received a previous treatment for their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Ability and willingness to comply with the requirements of the study protocol.
* Age ≥18 years.
* Have documented previously untreated chronic lymphocytic leukemia according to iwCLL / WHO criteria.
* Require treatment of CLL per iwCLL guidelines.
* CIRS score ≤ 6 (patient's CLL diagnosis is not included in CIRS score).
* Eastern Cooperative Oncology Group Performance Status of 0 or 1.
* Adequate hematologic function (unless caused by underlying disease, as established by extensive bone marrow involvement or as a result of hypersplenism secondary to the involvement of the spleen by CLL per the investigator) defined as follows:

  * Hemoglobin ≥ 8 g/dL without transfusion support, unless anemia is due to marrow involvement of CLL.
  * Absolute neutrophil count ≥ 1.0 x 10^9/L.
  * Platelet count ≥ 30 x 10^9/L; in cases of thrombocytopenia clearly due to marrow involvement of CLL (per the discretion of the investigator), platelet count should be ≥ 10 x 10^9/L if there is bone marrow involvement.
* Adequate renal function, as indicated by modified Cockcroft-Gault equation (eCCR; with the use of ideal body mass [IBM] instead of mass) of > 50mL/min
* Adequate liver function, as indicated by:

  * AST or ALT ≤ 2.5 x ULN.
  * Total bilirubin ≤ 1.5 x ULN (or ≤ 5 x ULN for patients with documented Gilbert syndrome).
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 30 days after the last dose of venetoclax or 18 months after the last dose of obinutuzumab, whichever is longer.

  * Women must refrain from donating eggs during this same period.
  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (> 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

  * With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 90 days after the last dose of venetoclax or 18 months after the last dose of obinutuzumab, whichever is longer. Men must refrain from donating sperm during this same period.
  * With pregnant female partners, men must remain abstinent or use a condom for the duration of the pregnancy to avoid exposing the embryo.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* Prior CLL-directed therapy. Patients may have received a brief (≤7 days) course of systemic steroids prior to initiation of study therapy for control of lymphoma-related symptoms.
* Transformation of CLL to aggressive NHL (Richter's transformation or prolymphocytic leukemia).
* Known hypersensitivity to any of the study drugs.
* History of prior malignancy, except for conditions as listed below if patients have recovered from the acute side effects incurred as a result of previous therapy:

  * Malignancies treated with curative intent and with no known active disease within 2 years
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease (no time constraint).
  * Adequately treated cervical carcinoma in situ without evidence of disease (no time constraint).
  * Surgically/adequately treated low grade, early stage, localized prostate cancer without evidence of disease (no time constraint).
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1 Day 1.
* Requires the use of warfarin (because of potential drug-drug interactions that may potentially increase the exposure of warfarin).
* Received the following agents within 7 days prior to the first dose of venetoclax:

  * Strong and moderate CYP3A inhibitors.
  * Strong and moderate CYP3A inducers.
  * Consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges), or star fruit within 3 days prior to the first dose of venetoclax.
* Clinically significant history of liver disease, including active viral or other hepatitis, current alcohol abuse, or cirrhosis
* Presence of positive test results for hepatitis B virus (HBV), hepatitis B surface antigen (HBsAg), or hepatitis C (HCV) antibody

  * Patients who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation
  * Patients with occult or prior HBV infection (defined as positive total hepatitis B core antibody [HBcAb] and negative HBsAg) may be included if HBV DNA is undetectable. These patients must be willing to undergo monthly DNA testing and should consider antiviral prophylaxis as per institutional standards.
* Known infection with HIV or human T-cell leukemia virus 1 (HTLV-1)
* Receipt of live-virus vaccines within 28 days prior to the initiation of study treatment or need for live-virus vaccines at any time during study treatment
* Pregnant or lactating, or intending to become pregnant during the study

  °Women of childbearing potential must have a negative serum pregnancy test result within 21 days prior to initiation of study drug per institutional standards.
* Recent major surgery (within 4 weeks prior to the start of Cycle 1, Day 1) other than for diagnosis.
* Inability to swallow a large number of tablets.
* Malabsorption syndrome or other condition that precludes enteral route of administration. This is subject to investigator discretion.
* Known allergy to both xanthine oxidase inhibitors and rasburicase.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 36 months

SECONDARY OUTCOMES:
Overall response rate | 2 years
  Overall response rate (ORR) is defined as the proportion of patients with a best overall response of partial response (PR) or complete response (CR). Patients who do not have a tumor response assessment for any reason will be considered non-responders and will be included in the denominator when calculating the ORR.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Thompson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Stanford University Medical Center (Data collection only), Stanford, California
  - Memorial Sloan Kettering Basking Ridge (All protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Commack (All protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Uniondale, New York
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm